CLINICAL TRIAL: NCT03901378
Title: A Phase II Trial of Pembrolizumab in Combination With Cisplatin or Carboplatin and Etoposide in Chemotherapy naïve Patients With Metastatic or Unresectable High Grade Gastroenteropancreatic or Lung (Excluding Small Cell) Neuroendocrine Carcinoma
Brief Title: Pembrolizumab With Chemotherapy in Metastatic or Unresectable High Grade Gastroenteropancreatic or Lung Neuroendocrine Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Ochsner Health System (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Robert Ramirez, Principal Investigator, Ochsner Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 55643/Pembrolizumab
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Neuroendocrine Carcinoma; Large Cell Neuroendocrine Carcinoma of the Lung; High Grade Neuroendocrine Carcinoma, Any Site
Keywords: Neuroendocrine carcinoma; Gastroenteropancreatic; Large cell neuroendocrine
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single Arm (Experimental): Pembrolizumab 200mg IV day 1 with Carboplatin AUC 6 IV day 1 or Cisplatin 80mg/m2 day 1 with etoposide 100mg/m2 days 1-3 of 21 day cycle. Repeat 4-6 cycles to be followed by maintenance Pembrolizumab 200mg IV day 1 every 21 days until progression or intolerance for up to 2 years.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Intravenous administration of pembrolizumab in combination with cisplatin or carboplatin and etoposide in first line metastatic or unresectable high grade neuroendocrine carcinoma:

SUMMARY:
The purpose of this study is to test the efficacy, safety, and tolerability of the combination of chemotherapy treatment, which could be either Cisplatin or carboplatin and etoposide, and the research study drug, Pembrolizumab (also known as MK-3475) in patients with high grade neuroendocrine carcinomas of the gastroenteropancreatic system or lung who are chemotherapy naïve. The chemotherapy treatment you receive will be either Cisplatin or carboplatin and etoposide. the participant's doctor will discuss this choice with you and determined which chemotherapy treatment is best for you.

DETAILED DESCRIPTION:
Combination chemotherapy is the mainstay of treatment for patients with high grade GEPNETs and neuroendocrine carcinomas of the lung.

This study will utilize pembrolizumab, a potent humanized immunoglobulin G4 (IgG4) monoclonal antibody (mAb) with high specificity of binding to the programmed cell death 1 (PD-1) receptor, thus blocks a protective mechanism of cancer cells and thereby allows the immune system to destroy them, in combination with chemotherapy.

Combination chemotherapy and pembrolizumab was recently FDA approved and ongoing trials are utilizing this or similar combination with preliminary data demonstrating a promising safety profile.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be 18 years of age on day of signing informed consent.
3. Must have cytologically or histologically proven high grade neuroendocrine carcinoma of the gastroenteropancreatic system or large cell neuroendocrine carcinoma as defined by the 2010 WHO classification.

   a. GEPNETs need to have Ki-67 greater than 55%.
4. Have metastatic or unresectable disease.
5. No prior systemic chemotherapy or immunotherapy for metastatic disease allowed.
6. Concurrent use of somatostatin analogs is allowed for symptom control.
7. Life expectancy greater than 12 weeks.
8. Have measurable disease based on RECIST 1.1.
9. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor/PI.
10. Have a performance status of 0 - 1 on the ECOG Performance Scale.
11. Demonstrate adequate organ function. All screening labs should be performed within 10 days of treatment initiation.
12. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
13. Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
14. Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
15. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had prior systemic anti-cancer therapy for metastatic or unresectable neuroendocrine tumors other than somatostatin analogs.
6. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
8. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
9. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
17. Has a known history of Human Immunodeficiency Virus (HIV).
18. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
19. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist) are live attenuated vaccines and are not allowed.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 1 year
  Assessed by investigator using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Combination therapy will be safe and tolerable compared to historical controls | Continuous from the signing of the informed consent to 28 days after last study treatment
  Collection of any adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ramirez, DO, Principal Investigator — Ochsneer Clinic Foudnation
Locations (2):
- United States (2):
  - Ochsner Clinic Foundation, Kenner, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No